CLINICAL TRIAL: NCT01130324
Title: VIBATIV (Telavancin Hydrochloride) Pregnancy Exposure Registry
Brief Title: VIBATIV Pregnancy Registry
Status: Withdrawn | Type: Observational
Why Stopped: Released by he FDA from this Post-Marketing Commitment
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 0113
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy
Keywords: VIBATIV; telavancin; Pregnancy; Registry
MeSH Terms: interventions — telavancin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VIBATIV treated pregnant women: Women treated with telavancin (any dose or duration) during pregnancy.
  Interventions: Drug: VIBATIV

INTERVENTIONS:
Drug: VIBATIV — Observational
  Other Names: telavancin; TD-6424

SUMMARY:
The purpose of this registry is to evaluate the outcome of pregnancy in women exposed to VIBATIV at any time during pregnancy. There are no mandated physician visits for the registry.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who were exposed to VIBATIV at any time during pregnancy
* Outcome of pregnancy is unknown at the time of enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to VIBATIV during pregnancy and where outcome of pregnancy is unknown at time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Outcomes of pregnancy in women exposed to VIBATIV at any time during pregnancy | Once per trimester, 6-7 months gestation, and within 4 weeks after the estimated due date

SECONDARY OUTCOMES:
Effect of fetal exposure to VIBATIV on pregnancy outcomes | Within 4 weeks after the estimated due date and if a live infant birth is reported, at 3, 6, 9, and 12 months of age.
Fetal/neonatal outcomes | Within 4 weeks after the estimated due date and if a live infant birth is reported, at 3, 6, 9, and 12 months of age.
Infant development and milestones through 12 months of age | Within 4 weeks after the estimated due date and if a live infant birth is reported, at 3, 6, 9, and 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Haberle, PhD, Principal Investigator — Cumberland Pharmaceuticals, Inc.
Locations (1):
- Cumberland Pharmaceuticals Inc., Nashville, Tennessee, United States